CLINICAL TRIAL: NCT03029910
Title: Eccentric Training and Cryotherapy Vs Eccentric Training and Whole Body Vibration in Achilles Tendinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Europea de Madrid (Other)
Responsible Party: Principal Investigator, Pedro Javier Martin, Principal Investigator, Universidad Europea de Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UEMadrid-Tendon01
Record Dates: First submitted 2017-01-17; First posted 2017-01-24 (Estimated); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Achilles Tendon; Tendinopathy
Keywords: Eccentric exercise; Whole body vibration; Cryotherapy
MeSH Terms: conditions — Tendinopathy | interventions — Cryotherapy; Vibration

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cryotherapy and eccentric exercise (Experimental)
  Interventions: Other: Cryotherapy and eccentric exercise
- Vibration and eccentric exercise (Experimental)
  Interventions: Other: Vibration and eccentric exercise
- Control (No Intervention)

INTERVENTIONS:
Other: Cryotherapy and eccentric exercise — 12 weeks, 5 days/week, once a day, 2 exercises, 3 sets/exercise, 15 repetition/set. Of excentric exercise of foot plantar flexors. First exercise with knee in extension. Second exercise with knee in flexion. Previously subjects should cool their leg in ice water during sixteen minutes at a temperature of 8ºC (+/-2ºC)
  Arms: Cryotherapy and eccentric exercise
Other: Vibration and eccentric exercise — 12 weeks, 5 days/week, once a day, 2 exercises, 3 sets/exercise, 15 repetition/set. Of excentric exercise of foot plantar flexors. First exercise with knee in extension. Second exercise with knee in flexion. During the exercise subjects will be subjected to vibration. Vibration parameters: Frequency: 35Hz, Amplitude: 4 millimeters, Force: 3,9G
  Arms: Vibration and eccentric exercise

SUMMARY:
The purpose of this study is to determine the effectiveness of eccentric exercise combined with vibration or cryotherapy in Achilles tendon pathology.

The investigators hypothesis is that the combined eccentric exercise is better than the results presented by the exclusive eccentric exercise.

This intervention differs from the classic studies in that we maintain the intensity throughout the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Sports people
* Positive initial ultrasound diagnosis
* Presence of degenerative changes at achilles mid portion
* Chronic Achilles tendon pain, (3/10 VAS)
* Pain when walking or running of Achilles tendon, (3/10 VAS)
* Pain in load in plantar flexion of Achilles tendon, 3/10 VAS)
* Pain in palpation of Achilles, (3/10 VAS)
* Morning Stiffness

Inclusion Criteria Healthy pople:

* Sports people
* Negative initial ultrasound diagnosis
* No syntomp of achilles tendinophaty

Exclusion Criteria:

* Receive physical, orthotic or physiotherapeutic treatment
* Asociated low back pain, ankle/knee/hip injury that may affect the study
* Previous injury or surgery of Achilles tendon.
* Pathologies that may limit the joint of ankle
* Pregnancy
* Obesity
* Patients with diabetes and/or other endocrine or metabolic pathologies or neurologic pathologies
* Patients diagnosed with cardiovascular disease
* Subjets diagnosed with familiar hypercholesterolemia and/or presence of xanthomas or with hyperuricemia
* Patients who have received renal transplantation
* Subjects who have suffered retinal detachment
* Subjects who have received oral contraceptives, statins, corticoids or hormone replacement therapy in the last six months
* Subjects who have received treatment wiht fluoroquinolones in the last two years
* Subjects who have received treatment with AINE's in the last four weeks

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2017-01-30 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2018-01-15 (Actual)

PRIMARY OUTCOMES:
Change at Achilles Tendon Cross Sectional Area | 3 months
  Ultrasound diagnosis.
Change at Achilles Tendon Thickness | 3 months
  Ultrasound diagnosis.

SECONDARY OUTCOMES:
Differences between healthy volunteers and volunteers with Achilles tendinopathy | 2 weeks
  Ultrasound diagnosis

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Europea, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No